CLINICAL TRIAL: NCT00243880
Title: SPOTRIAS: Neuroprotection With Statin Therapy for Acute Recovery Trial
Brief Title: Neuroprotection With Statin Therapy for Acute Recovery Trial (Neu-START)
Acronym: Neu-START
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Mitchell S Elkind, Associate Professor of Neurology and Epidemiology (in the Sergievsy Center), Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA5855; R01NS049060 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Stroke
Keywords: acute ischemic stroke; lovastatin; statin; neuroprotection; SPOTRIAS
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Lovastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lovastatin (Experimental): lovastatin at escalating dosages: 1 mg/kg/day, 3 mg/kg/day, 6 mg/kg/day, 8 mg/kg/day, 10 mg/kg/day
  Interventions: Drug: lovastatin

INTERVENTIONS:
Drug: lovastatin — investigators will treat the patients within 24 hours of symptom onset with short term high-dose lovastatin at escalating dosage. The escalating dosage levels will be 1, 3, 6, 8, and 10 mg/kg per day for 3 days.
  Other Names: Mevacor

SUMMARY:
The purpose of this dose escalation study is to evaluate the use of lovastatin for the treatment of acute ischemic stroke.

DETAILED DESCRIPTION:
The Neuroprotection with Statin Therapy for Acute Recovery Trial (Neu-START) is part of the Specialized Program on Translational Research in Acute Stroke (SPOTRIAS). The overall goals of SPOTRIAS are to enhance delivery of acute stroke patient care with a focus on high-risk, disadvantaged populations, train acute stroke translational researchers, and conduct 3 innovative acute stroke projects.

Neu-START will enroll 33 patients with acute ischemic stroke presenting within 24 hours of onset. In the trial, investigators will treat the patients within 24 hours of symptom onset with short term high-dose lovastatin at escalating dosage. The escalating dosage levels will be 1, 3, 6, 8, and 10 mg/kg per day for 3 days. Lovastatin is in a class of drugs called statins, used for lowering cholesterol and preventing cardiovascular disease. Patients will be followed for 30 days for clinical and laboratory outcome events.

The goals of this trial are to determine if lovastatin in increasing doses from 1 mg/kg to 10 mg/kg daily for 3 days beginning 24 hours after acute ischemic stroke can be administered safely, and to assess the pharmacokinetics of lovastatin administered at high doses.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Satisfies the criteria for ischemic stroke: acute focal neurological deficit of likely ischemic vascular origin.
* Patient or legally authorized representative has provided written informed consent prior to study entry.
* Patient can receive the first treatment dose within 0-24 hours of stroke onset. For patients found with stroke on awakening, it will be assumed that the stroke occurred the last time that the patient was known to be normal.
* Patient has pretreatment brain CT scan compatible with ischemic stroke and excludes hemorrhagic and non-vascular etiologies of symptoms.
* Patients taking statins at time of stroke may be included.

Exclusion Criteria:

* Brain imaging study shows a lesion other than ischemic stroke that could explain patient's symptoms (intracranial or subarachnoid hemorrhage, arteriovenous malformation, aneurysm, multiple sclerosis, tumor, abscess or other). Asymptomatic meningiomas are allowed.
* Patient had a stroke (ischemic or hemorrhagic) with residual deficit within 1 month prior to treatment.
* Mild stroke, defined as NIH Stroke Scale <2.
* Patient has received or is expected to receive intravenous rt-PA within 3 hours or intra-arterial rt-PA within 6 hours of stroke onset, according to our institutional standard of care.
* Receipt of intravenous rt-PA after 3 hours or intra-arterial rt-PA after 6 hours post-stroke onset.
* Seizure at presentation or within two weeks prior to stroke.
* Patient is comatose, regardless of etiology (> 4 points on the first three items of the NIHSS).
* History of intolerance or allergic reaction to any statins (myotoxicity, hepatic dysfunction, rash, etc.)
* Use of drugs within past 30 days that utilize the cytochrome CYP3A pathway (cyclosporine, itraconazole, ketoconazole, erythromycin, azithromycin, clarithromycin, nefazodone).
* Use of drugs within past 30 days that increase risk of myotoxicity with statins (gemfibrozil, other fibrates, niacin, amiodarone, verapamil).
* Baseline major electrolyte disturbances (sodium <125 or >150, potassium <3.0 or >5.5).
* Recent major trauma (<3 months).
* Hypothermia (body temperature < 96 degrees Fahrenheit).
* Baseline hypoxia (defined as oxygen saturation <92% on room air).
* History of likely or proven systemic viral infection within 30 days.
* Known HIV infection or use of protease inhibitors.
* Endocarditis likely as cause of stroke.
* Mitochondrial disorder likely as cause of stroke.
* Pregnancy or lactation.
* History of rhabdomyolysis, myopathy, or other severe muscle disease.
* History of hepatitis, decompensated liver disease (ascites, bleeding varices or encephalopathy), or liver failure.
* Liver function tests (ALT, AST) > 2X upper limit of normal.
* Unstable cardiovascular (includes uncontrolled hypertension), pulmonary, gastrointestinal, hepatic or musculoskeletal disease within one month (30 days) prior to treatment (by reported history).
* Patient has evidence of congestive heart failure or has history of end-stage cardiovascular disease (e.g. CHF NYHA Class III or IV or unstable angina).
* Abnormal ECG showing: Hemodynamically significant arrhythmia or frequent PVCs (>5/minute) (controlled atrial arrhythmia will not be an exclusion); evidence of acute myocardial infarction; Mobitz Type II 2nd degree AV block or 3rd degree AV block; ventricular tachycardia or ventricular fibrillation.
* Significant renal insufficiency, indicated by serum creatinine >2.0 mg/dl.
* Hypoglycemia (glucose < 60 mg/dl), significant hyperglycemia (glucose > 400 mg/dl) or diabetic ketoacidosis.
* Any of these hematologic abnormalities: Hb <10 g/dl; WBC <3.0 x 103/mm3; Platelet count <50,000/mm3
* Received an investigational drug within 30 days.
* Severe behavioral or social problems that may interfere with the conduct of clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
safety through 30 days defined as absence of liver or muscle-related toxicity on days 1, 2, 3, 5, 7, and 30. | 30 days
  Devt of clinical or laboratory evidence of major hepatic or muscle toxicity. Either: (1) liver toxicity: liver function test increase, devt jaundice, unexplained coagulopathy, or other clinical evidence of hepatitis or liver failure; or (2) muscle toxicity: increase in creatine phosphokinase (CK) at any time point

SECONDARY OUTCOMES:
pharmacokinetic measurements made on days 1, 3, 4, and 5. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Elkind, MD, MS, Principal Investigator — Columbia University; Ji Chong, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elkind MS, Sacco RL, MacArthur RB, Fink DJ, Peerschke E, Andrews H, Neils G, Stillman J, Corporan T, Leifer D, Cheung K. The Neuroprotection with Statin Therapy for Acute Recovery Trial (NeuSTART): an adaptive design phase I dose-escalation study of high-dose lovastatin in acute ischemic stroke. Int J Stroke. 2008 Aug;3(3):210-8. doi: 10.1111/j.1747-4949.2008.00200.x. PMID 18705902
- [Result] Elkind MS, Sacco RL, Macarthur RB, Peerschke E, Neils G, Andrews H, Stillman J, Corporan T, Leifer D, Liu R, Cheung K. High-dose lovastatin for acute ischemic stroke: results of the phase I dose escalation neuroprotection with statin therapy for acute recovery trial (NeuSTART). Cerebrovasc Dis. 2009;28(3):266-75. doi: 10.1159/000228709. Epub 2009 Jul 16. PMID 19609078